CLINICAL TRIAL: NCT05568277
Title: Evaluation of the Effectiveness of the Education Provided to Pregnant Women at Risk of Gestational Diabetes on Preventive Health Behaviors
Brief Title: Education of Pregnant Women at Risk of Gestational Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Burçin Bektaş Pardes, Research Assistant, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: bpardes1
Record Dates: First submitted 2022-09-25; First posted 2022-10-05 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2022-09

CONDITIONS: Pregnant Women; Gestational Diabetes
Keywords: pregnant women; gestational diabetes; Preventive Health; Education
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Intervention Model Description: intervention and control group
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education (Experimental): A minimum of 12-week training program and follow-up based on Pender's Health Promotion Model is planned until the 24th gestational week.
  Interventions: Behavioral: Education on preventive health behaviors based on Pender's Health Promotion Model
- Control (No Intervention): No intervention will be made by the researcher and they will receive routine antenatal care. After the post-test data are collected, the education booklet prepared by the researcher will be given to the pregnant women and sent to their e-mail addresses.

INTERVENTIONS:
Behavioral: Education on preventive health behaviors based on Pender's Health Promotion Model — Pregnant women included in the study will be given education on preventive health behaviors based on Pender's Health Promotion Model on the prevention of gestational diabetes over the web (ZOOM/Teams etc.) every two weeks. Pregnant women's questions will be answered. At the end of each training, data will be collected from pregnant women and follow-up charts will be filled. The education booklet prepared by the researcher will be given to the pregnant women after the first education and will be sent to their e-mail addresses.
  Arms: Education

SUMMARY:
There are studies in the literature showing that there is a decrease in the number of pregnant women diagnosed with gestational diabetes and improvements in parameters related to maternal and infant health, with the education to be given to pregnant women at risk of gestational diabetes on preventive lifestyle practices such as healthy nutrition, physical exercise, and coping with stress. The aim of this study; For pregnant women at risk of gestational diabetes; education on preventive health behaviors; It is to determine the level of knowledge about GDM, risk perception and its effect on healthy living behaviors.

DETAILED DESCRIPTION:
Gestational diabetes mellitus (GDM) is carbohydrate intolerance of varying degrees that begins during pregnancy or is first diagnosed during pregnancy. 4% of pregnancies are complicated by GDM. History of diabetes in first-degree relatives, history of GDM in previous pregnancies, body mass index over 30 kg/m2, significant weight gain during pregnancy, and maternal age over 25 are among the primary risk factors for gestational diabetes in pregnant women. Gestational diabetes; It causes serious maternal and fetal complications such as the risk of developing Type 2 diabetes in the mother, traumatic birth, preeclampsia, cesarean delivery, macrosomic baby, and congenital malformations.

It is known that healthy lifestyle behaviors are as effective as genetic factors in the development of diabetes. Lifestyle behavior modification is an essential component of gestational diabetes management. Studies show that 70-85% of pregnant women can control diabetes only with lifestyle changes. Protective health behaviors such as being at an ideal weight, eating healthy, exercising regularly and not smoking prevent the development of gestational diabetes. As a result of the Finnish Gestational Diabetes Prevention Study (RADIEL), it was found that physical activity and dietary intervention decreased the incidence of GDM by 36% in high-risk women. It is important that these preventive health behaviors are adopted and maintained by the pregnant woman. For this purpose, it is necessary to determine the problems in the process of acquiring behaviors that protect and improve health and prevent negative behaviors. Self-efficacy level plays an important role in initiating and maintaining preventive health behaviors. Education on preventive health behaviors can improve and improve self-care behaviors by increasing the self-efficacy level of women at risk of gestational diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Being between the 8th and 12th gestational weeks,
* Having risk factors for GDM (BMI of 30 kg/m2 and above, presence of diabetes in 1st degree relatives, diagnosis of GDM in previous pregnancy), being over 18 years old)
* Having a singleton pregnancy
* Ability to read and write Turkish
* Volunteering to participate in the study

Exclusion Criteria:

* Being older than 12 weeks of pregnancy
* Not having risk factors for GDM (BMI of 30 kg/m2 and above, presence of diabetes in 1st degree relatives, diagnosis of GDM in previous pregnancy), being over 18 years old)
* Having a multiple pregnancy
* Inability to read and write Turkish
* Not volunteering to participate in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women
Enrollment: 60 (Estimated)
Dates: Start 2023-04 (Estimated); Primary Completion 2023-04 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Pregnancy Physical Activity Questionnaire (PPAQ) | Baseline and between 30-32. gestational week
  The questionnaire, which determines the physical activity and exercise levels of pregnant women, consists of 35 questions. With this scale, housework and care activities of pregnant women (n=13), occupational activities (n=5), sports and exercise activities (n=8), transportation (n=3) and sedentary life (n=3) 32 activities are evaluated. The intensity of physical activity performed on the scale is expressed as MET (metabolic equivalent). When calculating the weekly energy expenditure of the activities, the time spent for each activity and the MET value of the activity are multiplied and the scores are expressed as MET hours per week (MET-hours/week). MET values vary according to the type of activity. Activity intensities are grouped as sedentary (<1.5 METs), mild (1.5-3.0 METs), moderate (3.0-6.0 METs), and severe (>0.6 METs). Following those calculations, women are classified as having a sedentary, light, moderate or severe physical activity levels.
Healthy Lifestyle Behaviours in Pregnancy Scale | Baseline and between 30-32. gestational week
  The Healthy Life Behaviors Scale in Pregnant Women is a five-point Likert-type scale filled in by the pregnant women themselves. The scale consists of a total of 29 items and 6 subscales: responsibility for pregnancy, hygiene, nutrition, physical activity, travel and acceptance of pregnancy. Each subscale of the scale can be used alone in studies. Scale items are scored from 5 to 1 from "always" to "never". There is no reverse entry item in the scale. High scores obtained from the scale indicate that pregnant women exhibit healthy lifestyle behaviors.
Pregnancy Risk Perception Questionnaire (PRPQ) | Baseline and between 30-32. gestational week
  It is a self-report questionnaire consisting of 9 visual analogue scales designed to measure a pregnant woman's perception of her pregnancy risks. This questionnaire consists of two subscales that include four questions about the risk to self (mother) and five questions about risk to the baby. Participants are asked to place a vertical mark on each item along a line giving a score between 0-100 to indicate their risk assessment. Total Pregnancy Risk Perception Questionnaire score is obtained by adding the score for each of the 9 items, and then dividing by 9. Higher scores indicate higher levels of perceived risk.
Diabetes Self-Efficacy Scale | between 30-32. gestational week
  The scale was developed to determine the self-efficacy of the patients with diabetes. The Likert-type scale consists of 8 items. The items of the scale are scored between 1 and 10 (1-Not at all confident, 10-Totally confident). The scale is usually applied within 5-6 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Gulten Guvenc, Study Director — Saglik Bilimleri Universitesi

IPD SHARING:
Plan to Share IPD: No
This study is planned as a doctoral dissertation.

REFERENCES:
- [Result] Rono K, Stach-Lempinen B, Eriksson JG, Poyhonen-Alho M, Klemetti MM, Roine RP, Huvinen E, Andersson S, Laivuori H, Valkama A, Meinila J, Kautiainen H, Tiitinen A, Koivusalo SB. Prevention of gestational diabetes with a prepregnancy lifestyle intervention - findings from a randomized controlled trial. Int J Womens Health. 2018 Aug 27;10:493-501. doi: 10.2147/IJWH.S162061. eCollection 2018. PMID 30214318
- [Result] Koivusalo SB, Rono K, Klemetti MM, Roine RP, Lindstrom J, Erkkola M, Kaaja RJ, Poyhonen-Alho M, Tiitinen A, Huvinen E, Andersson S, Laivuori H, Valkama A, Meinila J, Kautiainen H, Eriksson JG, Stach-Lempinen B. Gestational Diabetes Mellitus Can Be Prevented by Lifestyle Intervention: The Finnish Gestational Diabetes Prevention Study (RADIEL): A Randomized Controlled Trial. Diabetes Care. 2016 Jan;39(1):24-30. doi: 10.2337/dc15-0511. Epub 2015 Jul 29. PMID 26223239
- [Result] Chasan-Taber L. Lifestyle interventions to reduce risk of diabetes among women with prior gestational diabetes mellitus. Best Pract Res Clin Obstet Gynaecol. 2015 Jan;29(1):110-22. doi: 10.1016/j.bpobgyn.2014.04.019. Epub 2014 Aug 19. PMID 25220104